CLINICAL TRIAL: NCT02550873
Title: A Phase 2 Trial to Evaluate the Efficacy of PRM-151 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Trial to Evaluate the Efficacy of PRM-151 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA42404; PRM-151-202 (Other: Promedior, Inc.); 2014-004782-24 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-16 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — PRM-151

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRM-151 10mg / kg (Experimental): Dosing Every 4 Weeks
  Interventions: Biological: PRM-151
- Placebo (Placebo Comparator): Dosing Every 4 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Biological: PRM-151 — PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
  Arms: PRM-151 10mg / kg
Other: placebo — Placebo IV infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks
  Arms: Placebo

SUMMARY:
This study is a Phase 2, randomized, double-blind, placebo controlled, pilot study designed to evaluate the efficacy and safety of PRM-151 administered through Week 24 to subjects with IPF.

DETAILED DESCRIPTION:
PRM-151 is an anti-fibrotic immunomodulator being developed for treatment of fibrotic diseases.

ELIGIBILITY:
Inclusion Criteria

1. Is aged 40-80 years.
2. Has IPF satisfying the American Thoracic Society/European Respiratory Society /Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) diagnostic criteria (Raghu, Collard et al. 2011). In the absence of a surgical lung biopsy, high-resolution computed tomography (HRCT) must be "consistent with "usual interstitial pneumonia" (UIP) defined as meeting either criteria A, B, and C, or criteria A and C, or criteria B and C below:

   * Definite honeycomb lung destruction with basal and peripheral predominance.
   * Presence of reticular abnormality AND traction bronchiectasis consistent with fibrosis, with basal and peripheral predominance.
   * Atypical features are absent, specifically nodules and consolidation. Ground glass opacity, if present, is less extensive than reticular opacity pattern.
3. If on pirfenidone or nintedanib, subject must have been on a stable dose of pirfenidone or nintedanib for at least 3 months without increase in forced vital capacity (FVC)% predicted on two consecutive pulmonary function tests (PFTs), including screening PFTs. Subjects may not be on both pirfenidone and nintedanib.
4. If not currently receiving pirfenidone or nintedanib, subject must have been off pirfenidone or nintedanib for ≥ 4 weeks before baseline.
5. Has a FVC ≥ 50% and ≤ 90% of predicted.
6. Has a DLCO ≥ 25% and ≤ 90% of predicted.
7. Minimum distance on 6-Minute Walk Test (6MWT) of 150 meters.
8. Has a forced expiratory volume in 1 second (FEV1)/FVC ratio > 0.70.
9. Women of child bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤ 55 years or 12 months if > 55 years, must have a negative serum pregnancy test within four weeks prior to the first dose of study drug and must agree to use adequate methods of birth control throughout the study. Adequate methods of contraception are defined in the protocol.
10. Has a life expectancy of at least 9 months
11. According to the investigator's best judgment, can comply with the requirements of the protocol.
12. Has provided written informed consent to participate in the study.

Exclusion Criteria:

1. Has emphysema ≥ 50% on HRCT or the extent of emphysema is greater than the extent of fibrosis according to reported results from the most recent HRCT.
2. Has a history of cigarette smoking within the previous 3 months.
3. Has received investigational therapy for IPF within 4 weeks before baseline.
4. Is receiving systemic corticosteroids equivalent to prednisone > 10 mg/day or equivalent within 2 weeks of baseline.
5. Received azathioprine, cyclophosphamide, or cyclosporine A within 4 weeks of baseline.
6. Has a history of a malignancy within the previous 5 years, with the exception of basal cell skin neoplasms. In addition, a malignant diagnosis or condition first occurring prior to 5 years must be considered cured, inactive, and not under current treatment.
7. Has any concurrent condition other than IPF that, in the Investigator's opinion, is unstable and/or would impact the likelihood of survival for the study duration or the subject's ability to complete the study as designed, or may influence any of the safety or efficacy assessments included in the study.
8. Has baseline resting oxygen saturation of < 89% on room air or supplemental oxygen.
9. Is unable to refrain from use of the following:

   * Short acting bronchodilators on the day of and within 12 hours of pulmonary function, DLCO, and 6 minute walk assessments.
   * Long acting bronchodilators on the day of and within 24 hours of these assessments.
10. Has a known post bronchodilator (short acting beta agonist [SABA] - albuterol or salbutamol) increase in FEV1 of >10% and in FVC of >7.5%.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernt van den Blink, MD, PhD, Study Director — Hoffmann-La Roche
Locations (18):
- United States (10):
  - UCSF Interstitial Lung Disease Program, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - UT - Southwestern Medical School, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- Thomayer Hospital, Prague, Czechia
- Germany (2):
  - Justus-Liebig University Giessen, Giessen
  - Thoraxklinik University of Heidelberg, Heidelberg
- Italy (2):
  - Az. Ospedaliera Universitaria-Policlinico V. Emanuele di Catania, Catania
  - Azienda Ospedaliera San Gerardo, Monza
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Hospital University de Bellvitge, Barcelona, Spain
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland

REFERENCES:
- [Result] Raghu G, van den Blink B, Hamblin MJ, Brown AW, Golden JA, Ho LA, Wijsenbeek MS, Vasakova M, Pesci A, Antin-Ozerkis DE, Meyer KC, Kreuter M, Santin-Janin H, Mulder GJ, Bartholmai B, Gupta R, Richeldi L. Effect of Recombinant Human Pentraxin 2 vs Placebo on Change in Forced Vital Capacity in Patients With Idiopathic Pulmonary Fibrosis: A Randomized Clinical Trial. JAMA. 2018 Jun 12;319(22):2299-2307. doi: 10.1001/jama.2018.6129. PMID 29800034
- [Derived] Raghu G, Hamblin MJ, Brown AW, Golden JA, Ho LA, Wijsenbeek MS, Vasakova M, Pesci A, Antin-Ozerkis DE, Meyer KC, Kreuter M, Burgess T, Kamath N, Donaldson F, Richeldi L. Long-term evaluation of the safety and efficacy of recombinant human pentraxin-2 (rhPTX-2) in patients with idiopathic pulmonary fibrosis (IPF): an open-label extension study. Respir Res. 2022 May 21;23(1):129. doi: 10.1186/s12931-022-02047-0. PMID 35597980
- [Derived] Raghu G, van den Blink B, Hamblin MJ, Brown AW, Golden JA, Ho LA, Wijsenbeek MS, Vasakova M, Pesci A, Antin-Ozerkis DE, Meyer KC, Kreuter M, Moran D, Santin-Janin H, Aubin F, Mulder GJ, Gupta R, Richeldi L. Long-term treatment with recombinant human pentraxin 2 protein in patients with idiopathic pulmonary fibrosis: an open-label extension study. Lancet Respir Med. 2019 Aug;7(8):657-664. doi: 10.1016/S2213-2600(19)30172-9. Epub 2019 May 20. PMID 31122893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred fifty-one (151) patients were screened for the study. Of these, one hundred seventeen (117) were found to be eligible and were randomized. One randomized patient dropped out of the study prior to receiving any study drug.
Groups:
- PRM-151 10 mg/kg; Open Label PRM-151 10 mg/kg: Dosing Every 4 Weeks
  PRM-151: PRM-151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
Period: Randomized Double Blind
Arm/Group | PRM-151 10 mg/kg | Placebo | Open Label PRM-151 10 mg/kg
Started (Number of patients randomized) | 78 | 39 | 0
Received Treatment | 77 | 39 | 0
Continue to Open Label Extension | 74 | 37 | 0
Completed | 74 | 37 | 0
Not Completed | 4 | 2 | 0
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Disease progression | 1 | 1 | 0
Period: Open Label Extension
Arm/Group | PRM-151 10 mg/kg | Placebo | Open Label PRM-151 10 mg/kg
Started | 0 | 0 | 111
Completed | 0 | 0 | 0 (Open Label extension is ongoing)
Not Completed | 0 | 0 | 111
Not completed — Study ongoing | 0 | 0 | 111

BASELINE CHARACTERISTICS:
Population: All treated patients
Groups:
- PRM-151 10 mg/kg: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
- Total: Total of all reporting groups
Arm/Group | PRM-151 10 mg/kg | Placebo | Total
Number analyzed (Participants) | 77 | 39 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 14 | 38
  >=65 years | 53 | 25 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 65 | 29 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: White | 74 | 39 | 113
  Ethnicity/Race: Black/African | 1 | 0 | 1
  Ethnicity/Race: Hispanic | 1 | 0 | 1
  Ethnicity/Race: Asian | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 86.1 (15.2) | 87.5 (13.4) | 86.5 (14.5)
Years since IPF diagnosis, mean (SD) [Mean (Standard Deviation); unit: years] | 3.74 (2.16) | 3.90 (2.62) | 3.79 (2.32)
FVC [Mean (Standard Deviation); unit: mL] | 2733 (630) | 2763 (654) | 2743 (635)
FVC [% predicted] [Mean (Standard Deviation); unit: Percentage of predicted FVC] | 67.7 (10.9) | 67.4 (11.4) | 67.6 (11.0)
FEV1/FVC [Mean (Standard Deviation); unit: Percentage of FEV1/FVC] | 81.2 (5.1) | 81.6 (4.7) | 81.3 (4.9)
Hemoglobin-corrected DLCO [Mean (Standard Deviation); unit: Percentage of predicted DLCO] | 40.1 (9.1) | 43.2 (10.5) | 41.2 (9.7)
6MWD [Median (Standard Deviation); unit: meters] | 434.8 (92.5) | 457.7 (117.7) | 442.5 (101.7)
SpO2 at rest [Mean (Standard Deviation); unit: Percentage of SpO2] | 95.6 (2.1) | 95.5 (1.8) | 95.6 (2.0)
IPF Therapy Status at Baseline [Count of Participants; unit: Participants]
  Concurrent IPF Therapy | 61 | 30 | 91
  Concurrent pirfenidone | 39 | 22 | 61
  Concurrent nintedanib | 22 | 8 | 30
  No concurrent IPF therapy | 16 | 9 | 25
  IPF therapy naiive | 8 | 7 | 15
Comorbid Conditions [Count of Participants; unit: Participants]
  GERD | 47 | 16 | 63
  Hypertension | 38 | 14 | 52
  Cardiac Disorders | 29 | 7 | 36
  Coronary Artery Disorders | 15 | 4 | 19
  Emphysema | 2 | 0 | 2
  Pulmonary Hypertension | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) [% Predicted]
Description: Determine the effect size of PRM-151 relative to placebo in change from Baseline to Week 28 in mean FVC% predicted, pooling subjects on a stable dose of pirfenidone or nintedanib with subjects not on other treatment for IPF.
Time Frame: 0 to 28 weeks
Population: All treated patients
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of predicted FVC
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Percentage of predicted FVC | -2.5 [-3.2 to -1.8] | -4.8 [-5.7 to -3.8]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg vs Placebo; The sample size calculation was based on the following assumptions: Normal distribution Homogeneity of variance the same in both arms, and for both types of patients Randomization ratio PRM-151:placebo = 2:1 Expected value for patients on pirfenidone or nintedanib = -1.5 Expected value for patients on no other treatment = -3 Expected value for patients on PRM-151 ≥ 0.75 Standard deviation = 5 75% of patients on a stable dose of pirfenidone or nintedanib α=0.10 two-sided Power = 80%; Test type: Superiority; p = 0.0014, Mixed Models Analysis — a priori threshold for statistical significance = 0.10; Random intercept; dependent variable=raw values at each time point; explanatory variables=stratum, treatment, time and treatment by time interaction; Mean Difference (Net) = 2.3, 90% CI 2-sided [1.1 to 3.5], Standard Error of Mean 0.72

2. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD)
Time Frame: 0 to 28 weeks
Population: All treated patients
Measure: Least Squares Mean (90% Confidence Interval); unit: meters
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
meters | -0.5 [-8.6 to 7.6] | -31.8 [-43.0 to -20.5]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis — This study was not powered to test hypothesis beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 31.3, 90% CI 2-sided [17.4 to 45.1], Standard Error of Mean 8.42

3. Secondary Outcome: Change From Baseline in Total Lung Volume on High-resolution Computed Tomography (HRCT)
Description: Mean change from baseline in total lung volume on HRCT using quantitative imaging software.
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had HRCT data at both the Baseline and Week 28 time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliliters
Groups:
- PRM-151 10 mg/kg; No Background Therapy: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks in patients not receiving concurrent pirfenidone or nintedanib
- PRM-151 10 mg/kg; Pirfenidone or Nintedanib: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks in patients receiving concurrent pirfenidone or nintedanib
- Placebo; No Background Therapy: Dosing Every 4 weeks
  placebo: Placebo IV infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks in patients not receiving concurrent pirfenidone or nintedanib
- Placebo; Pirfenidone or Nintedanib: Dosing Every 4 weeks
  placebo: Placebo IV infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks in patients receiving concurrent pirfenidone or nintedanib
Arm/Group | PRM-151 10 mg/kg; No Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo; No Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 14 | 52 | 8 | 26
milliliters | -103.8 [-234.1 to 26.6] | -108.1 [-184.2 to -31.9] | -197.3 [-341.2 to -53.3] | -201.6 [-305.3 to -97.9]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg; No Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo; No Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.2032, Mixed Models Analysis — This study was not powered to test hypothesis beyond the primary endpoint; Random intercept and slope; dependent variable=raw values; explanatory variables=stratum, treatment, time and treatment by time interaction; Mean Difference (Net) = 93.5, 90% CI 2-sided [-27.7 to 214.7], Standard Error of Mean 72.98

4. Secondary Outcome: Change From Baseline in Volume of Interstitial Lung Abnormalities (ILA) on HRCT
Description: Mean change from baseline in volume of parenchymal features on HRCT representative of ILA, including ground glass density, reticular changes, and honeycombing, using quantitative imaging software
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had HRCT data at both the Baseline and Week 28 time points.
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | PRM-151 10 mg/kg; No Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo; No Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 14 | 52 | 8 | 26
milliliters | 49.7 (49.65) | 80.9 (29.21) | 17.8 (55.26) | 49.0 (39.64)
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg; No Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo; No Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.4927, Mixed Models Analysis — This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 31.9, 90% CI 2-sided [-45.0 to 108.8], Standard Error of Mean 46.33

5. Secondary Outcome: Change From Baseline in % of Total Lung Volume of ILA on HRCT
Description: Mean change from baseline in % of total lung volume of parenchymal features on HRCT representative of ILA, including ground glass density, reticular changes, and honeycombing, using quantitative imaging software
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had HRCT data at both the Baseline and Week 28 time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of total lung volume
Groups:
- PRM-151 10 mg/kg, no Background Therapy: Dosing Every 4 Weeks
  PRM-151: PRM-151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
- PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib; Placebo, no Background Therapy; Placebo; Pirfenidone or Nintedanib: Dosing Every 4 weeks
  placebo: Placebo IV infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 14 | 52 | 8 | 26
percentage of total lung volume | 2.6 [-0.9 to 6.0] | 3.0 [1.0 to 5.1] | 1.5 [-2.4 to 5.4] | 1.9 [-0.8 to 4.7]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.5835, Mixed Models Analysis — This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.1, 90% CI 2-sided [-2.2 to 4.3], Standard Error of Mean 1.96

6. Secondary Outcome: Change From Baseline in Volume of Normal Lung on HRCT
Description: Mean change from baseline in volume of parenchymal features on HRCT representative of normal lung (non-ILA), including normal and mild low attenuation areas, using quantitative imaging software.
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had HRCT data at both the Baseline and Week 28 time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliliters
Groups:
- PRM-151 10 mg/kg; Pirfenidone or Nintedanib: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks in patients receiving concurrent pirfenidone or nintedanib therapy
- Placebo; Pirfenidone or Nintedanib: Dosing Every 4 weeks
  placebo: Placebo IV infusion over 60 minutes on days 1, 3, and 5, then one infusion every 4 weeks in patients not receiving concurrent pirfenidone or nintedanib
Arm/Group | PRM-151 10 mg/kg; No Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo; No Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 14 | 52 | 8 | 26
milliliters | -165.2 [-347.2 to 16.8] | -201.1 [-307.6 to -94.5] | -208.8 [-410.1 to -7.5] | -244.7 [-389.9 to -99.4]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg; No Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo; No Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.6707, Mixed Models Analysis — This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 43.6, 90% CI 2-sided [-126.3 to 213.5], Standard Error of Mean 102.28

7. Secondary Outcome: Change From Baseline in % of Normal Lung on HRCT (%)
Description: Mean change from baseline in % of total lung volume of parenchymal features on HRCT representative of normal lung (non-ILA), including normal and mild low attenuation areas, using quantitative imaging software.
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had HRCT data at both the Baseline and Week 28 time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of total lung volume
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 14 | 52 | 8 | 26
percentage of total lung volume | -2.6 [-6.0 to 0.8] | -3.3 [-5.3 to -1.3] | -1.4 [-5.1 to 2.4] | -2.1 [-4.8 to 0.7]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.52, Mixed Models Analysis — This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.2, 90% CI 2-sided [-4.4 to 1.9], Standard Error of Mean 1.91

8. Secondary Outcome: Correlation Between Mean Change From Baseline in FVC [% Predicted] and Mean Change From Baseline in ILA
Description: Correlation between mean change from Baseline in FVC [% predicted] and mean change from Baseline in volume of parenchymal features on HRCT representative of ILA, including ground glass density, reticular changes, and honeycombing by quantitative imaging software.
Time Frame: 0 to 28 weeks
Population: All patients from the ATS population who had FVC and HRCT data at both the Baseline and Week 28 time points.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 60 | 33
Correlation coefficient | -0.5027 [-0.6686 to -0.2812] | -0.4570 [-0.6880 to -0.1279]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg; Test type: Other — Correlation analysis; p = 0.0001, Pearson's correlation — This study was not powered to test hypotheses beyond the primary endpoint
Statistical Analysis 2: Comparison: Placebo; This study was not powered to test hypotheses beyond the primary endpoint; Test type: Other — Correlation analysis; p = 0.0069, Pearson's correlation

9. Secondary Outcome: Number of Subjects With a Decline in FVC [% Predicted] of ≥ 5% and ≥ 10% From Baseline to Week 28.
Description: Pulmonary Function Tests for the Proportion (%) of subjects with a decline in FVC% predicted of ≥ 5% and ≥ 10% from Baseline to Week 28.
Time Frame: 0 to 28 weeks
Population: All treated patients with data at baseline and 28 weeks
Measure: Count of Participants; unit: Participants
Groups:
- PRM-151 10 mg/kg, no Background Therapy; PRM-151 10 mg/kg; Pirfenidone or Nintedanib; Placebo; Pirfenidone or Nintedanib: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 13 | 54 | 8 | 27
Participants
  Decline in % Predicted FVC ≥ 5% | 2 | 18 | 2 | 11
  Decline in % Predicted FVC ≥10% | 1 | 1 | 0 | 3
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.4179, Mixed Models Analysis — P-Value for decline in % Predicted FVC ≥ 5%. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.2184, Mixed Models Analysis — P-Value for decline in % predicted FVC ≥ 10%. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Subjects With a Decline in FVC of ≥ 100 mL and ≥ 200 mL From Baseline to Week 28.
Time Frame: 0 to 28 weeks
Population: All treated patients with data at baseline and Week 28
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 13 | 54 | 8 | 27
Participants
  Decrease in FVC ≥ 100 mL | 5 | 32 | 2 | 16
  Decrease in FVC ≥ 200 mL | 2 | 19 | 1 | 8
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.7773, Mixed Models Analysis — P-Value for decline in FVC ≥ 100 mL. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.5976, Mixed Models Analysis — P-Value for decline in FVC ≥ 200 mL. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Subjects With an Increase in FVC [% Predicted] of ≥ 5% and ≥10% From Baseline to Week 28.
Time Frame: 0 to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 16 | 61 | 9 | 30
Participants
  Increase in % Predicted FVC ≥5% | 1 | 1 | 0 | 0
  Increase in % Predicted FVC ≥10% | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.29, Mixed Models Analysis — P-Value for increase in % predicted FVC ≥ 5%. P-Value for an increase in % predicted FVC ≥ 10% not reported. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Subjects With an Increase in FVC of ≥ 100 mL and ≥ 200 mL From Baseline to Week 28
Time Frame: 0 to 28 weeks
Population: All treated patients with FVC data at Baseline and Week 28
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 13 | 54 | 8 | 27
Participants
  Increase in FVC ≥ 100 mL | 1 | 6 | 0 | 0
  Increase in FVC ≥ 200 mL | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.0508, Mixed Models Analysis — P-Value for increase in FVC ≥ 100 mL. P-Value for increase in FVC ≥ 200 mL not reported. This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

13. Secondary Outcome: Number of Subjects With Stable Disease, Defined as a Change in FVC [% Predicted] of < 5% From Baseline to Week 28.
Time Frame: 0 to 28 weeks
Population: All treated subjects with data at baseline and week 28
Measure: Count of Participants; unit: Participants
Groups:
- PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib; Placebo; Pirfenidone or Nintedanib: Dosing Every 4 Weeks
  PRM-151: PRM 151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 13 | 54 | 8 | 27
Participants | 10 | 35 | 6 | 16
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.6308, Mixed Models Analysis — This study was not powered to test hypotheses beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

14. Secondary Outcome: Number of Subjects With Stable Disease, Defined as a Change in FVC of < 100 mL From Baseline to Week 28.
Time Frame: 0 to 28 weeks
Population: All treated subjects with FVC data at Baseline and Week 28
Measure: Count of Participants; unit: Participants
Groups:
- PRM-151 10 mg/kg; Pirfenidone or Nintedanib: Dosing Every 4 weeks
  PRM-151: PRM-151 10 mg/kg IV infusion over 60 minutes days 1, 3, and 5, then one infusion every 4 weeks
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 13 | 54 | 8 | 27
Participants | 7 | 16 | 6 | 11
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.1846, Mixed Models Analysis — This study was not powered to test hypothesis beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]

15. Secondary Outcome: Change From Baseline in % Predicted Diffusion Capacity of Carbon Monoxide (DLCO).
Description: Pulmonary Function Tests to discern the mean change from Baseline to Week 28 in % predicted diffusion capacity of carbon monoxide (DLCO).
Time Frame: 0 to 28 weeks
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of predicted DLCO
Arm/Group | PRM-151 10 mg/kg, no Background Therapy | PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib | Placebo, no Background Therapy | Placebo; Pirfenidone or Nintedanib
Number analyzed (Participants) | 16 | 61 | 9 | 30
percentage of predicted DLCO | -2.8 [-5.1 to -0.5] | -3.0 [-4.4 to -1.6] | -2.4 [-5.0 to 0.3] | -2.5 [-4.4 to -0.7]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg, no Background Therapy vs PRM-151 10 mg/kg IV; Pirfenidone or Nintedanib vs Placebo, no Background Therapy vs Placebo; Pirfenidone or Nintedanib; Test type: Superiority; p = 0.7424, Mixed Models Analysis — This study was not powered to test hypothesis beyond the primary endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.4, 90% CI 2-sided [-2.6 to 1.7], Standard Error of Mean 1.31

16. Secondary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Tolerability/safety was assessed over the 28-week study period by the number of reported TEAEs
Time Frame: 0 to 28 weeks
Population: Safety population (All randomized patients who received at least one dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 71 | 36

17. Secondary Outcome: Percentage of Subjects Discontinuing Study Drug Due to AEs
Description: Tolerability/safety was assessed over the 28-week study period by the proportion of subjects who discontinued study drug due to AEs
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 2 | 1

18. Secondary Outcome: Percentage of Subjects Reporting Serious Adverse Events (SAEs)
Description: Tolerability/safety was assessed over the 28-week study period by incidence of SAEs
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 6 | 4

19. Secondary Outcome: Percentage of Subjects Reporting Respiratory Decline AEs
Description: Tolerability/safety was assessed over the 28-week study period by the number of reported respiratory decline AEs, defined as follows:
  * Unscheduled visits to a healthcare professional for respiratory status deterioration.
  * Urgent care visits for respiratory status deterioration.
  * Hospitalization due to a worsening or exacerbation of respiratory symptoms.
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 11 | 4

20. Secondary Outcome: Percentage of Subjects Reporting Respiratory Decline SAEs [Safety and Tolerability]
Description: Tolerability/safety was assessed over the 28-week study period by the number of reported serious respiratory decline AEs
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 4 | 4

21. Secondary Outcome: Percentage of Subjects With Infusion Related Reactions
Description: Infusion Related Reactions were defined as events of headache, fever, facial flushing, pruritus, myalgia, nausea, chest tightness, dyspnea, vomiting, erythema, abdominal discomfort, diaphoresis, shivers, hypertension, hypotension, lightheadedness, palpitations, urticaria and somnolence occurring between the start of a study treatment infusion and one hour after completion of the infusion.
Time Frame: 0 to 28 weeks
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants
  Any Infusion Related Reaction | 2 | 1
  Dizziness | 1 | 0
  Hypertensive crisis | 1 | 1

22. Secondary Outcome: All Cause Mortality
Description: Tolerability/safety was assessed over the 28-week study period by the incidence of all cause mortality
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 0 | 1

23. Secondary Outcome: Mortality Due to Respiratory Deterioration
Description: Tolerability/safety was assessed over the 28-week study period by the incidence of mortality due to respiratory deterioration
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 0 | 1

24. Secondary Outcome: Mortality Due to Disease Related Events
Description: Number of patients who died over the 28 week study period due to disease-related events (defined as cough, IPF exacerbation, IPF progression and respiratory decline AEs)
Time Frame: 0 to 28 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
Participants | 0 | 0

25. Other Pre Specified Outcome: Change From Baseline in FVC Volume
Time Frame: 0 to 28 weeks
Population: All treated subjects
Measure: Least Squares Mean (90% Confidence Interval); unit: milliliters
Arm/Group | PRM-151 10 mg/kg | Placebo
Number analyzed (Participants) | 77 | 39
milliliters | -127.7 [-181.8 to -73.5] | -242.3 [-317.2 to -167.3]
Statistical Analysis 1: Comparison: PRM-151 10 mg/kg vs Placebo; Test type: Superiority; p = 0.0416, Mixed Models Analysis — This study was not powered to test hypothesis beyond the primary endpoint; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 114.6, 90% CI 2-sided [22.2 to 207.1], Standard Deviation 56.10

ADVERSE EVENTS:
Time Frame: 28 Weeks
Arm/Group | PRM-151 10 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 1/39
Serious Adverse Events (participants affected / at risk) | 6/77 | 4/39
Other Adverse Events (participants affected / at risk) | 58/77 | 28/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRM-151 10 mg/kg (N=77) | Placebo (N=39)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRM-151 10 mg/kg (N=77) | Placebo (N=39)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 2 (2)
Fatigue (General disorders) | 13 (20) | 4 (4)
Nasopharyngitis (Infections and infestations) | 12 (15) | 9 (13)
Headache (Nervous system disorders) | 11 (15) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 2 (2)
Bronchitis (Infections and infestations) | 8 (8) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (8)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 4 (5) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 3 (4)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Dizziness (Nervous system disorders) | 6 (7) | 3 (4)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (5)
Influenza-like illness (General disorders) | 3 (4) | 2 (5)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (8)
Depression (Psychiatric disorders) | 0 (0) | 2 (5)

LIMITATIONS AND CAVEATS:
Study not designed to test secondary outcome measures. Diagnosis of IPF allowed "possible usual interstitial pneumonia." HRCTs read locally, so reads may be heterogeneous. HRCTs are susceptible to inspiratory effort artifacts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A Publications Committee comprised of Investigators participating in the study and representatives from Promedior was formed to oversee the publication of the study results, which reflected the experience of all participating study centers. Subsequently, individual Investigators may publish results from the study in compliance with their agreement with the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT02550873/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02550873/SAP_003.pdf